CLINICAL TRIAL: NCT05870059
Title: Comparative Evaluation of Propolis Mouthwash With 0.2% Chlorhexidine Mouthwash in Improving the Periodontitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Dr. Maliha Waqar, Principal Investigstor, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4300921MWOM
Record Dates: First submitted 2023-04-11; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: As this is going to be a double-blind study, a third person will dispense the Propolis mouthwash (prepared in Ziauddin College of pharmacy) and Chlorhexidine mouthwash (commercially available) into dark-colored bottles of the same size and shape. The third person will code the bottles as A or B and seal the codes with the product name in envelopes accordingly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propolis (Experimental): 5 ml of 20% propolis mouthwash twice a day.
  Interventions: Drug: Propolis mouthwash
- chlorhexidine (Active Comparator): 5 ml of 0.2% chlorhexidine mouthwash twice a day.
  Interventions: Drug: Chlorhexidine mouthwash

INTERVENTIONS:
Drug: Propolis mouthwash — After scaling and root planning at the baseline visit, patients were prescribed to use 5ml of propolis mouthwash twice a day for 6 weeks. patients were also prescribed to not eat and drink anything for half an hour after the rinse.
  Arms: propolis
Drug: Chlorhexidine mouthwash — After scaling and root planning at the baseline visit, patients were prescribed to use chlorhexidine mouthwash twice a day for 6 weeks. patients were also prescribed to not eat and drink anything for half an hour after the rinse.
  Other Names: clinica mouthwash
  Arms: chlorhexidine

SUMMARY:
The goal of this clinical trial is to compare the efficacy of Propolis mouthwash with 0.2% Chlorhexidine mouthwash as an adjunct to mechanical therapy in improving the status of periodontal disease in peri-menopausal women.

The main question it aims to answer are:

* Will propolis mouthwash be equal to Chlorhexidine mouthwash in improving the periodontal status of perimenopausal women?
* Can neopterin be used as an indicator of periodontal disease.

Participants will be asked questions about their general health, menstrual health and oral health then scaling will be done. After that participants will give saliva sample by spitting in a given container. Participants will be divided into 2 groups for treatment and each group comprised of 51 participants.

Group 1: 20% Propolis mouthwash, twice a day for 6 weeks. Group 2: 0.2% chlorhexidine mouthwash, twice a day for 6 weeks.

DETAILED DESCRIPTION:
Patients who gave consent underwent oral examination and subjects with scores 3 and 4 according to the protocols described by the British Society of Periodontology were recruited into the study.

To evaluate the treatment outcome following periodontal parameters were assessed at baseline, 6 weeks and 12 weeks.

a) periodontal pocket depth b) clinical attachment loss c) bleeding on probing.

The development of mouthwash includes 2 steps i.e. extraction and formulation. i) Propolis extraction was carried out at the University of Karachi, and the propolis collected was authenticated by the Department of Pharmacognosy, Faculty of Pharmacy, University of Karachi.

ii) The formulation was done by the Department of Pharmacognosy at Ziauddin College of Pharmacology.

After formulations, various stability tests were performed on mouthwash to check its safety such as pH, Viscosity, Bio-burden and skin irritancy test. In the end, participants were also asked questions to check the acceptability of the product in terms of odour, colour, taste, fragrance, application and satisfaction with the outcome by the participants. those items that achieved acceptance of 80% or above were considered acceptable.

Saliva samples were taken at baseline and 12 weeks and neopterin levels were assessed using ELISA.

The correlation between neopterin levels and measures of clinical parameters after the treatment is made to evaluate if neopterin can be used as an indicator of disease progression and treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Females of age 40-50 years.
* Patients who are willing to receive treatment and give informed consent.
* Patients with probing pocket depth (PPD) of 4mm - 5mm and clinical attachment loss (CAL) of 1-4 mm.
* Presence of bleeding on probing (BOP).
* Patients should not have been subject to periodontal therapy and antibiotic medication in the past 6 months.
* Patients with a minimum of 20 teeth in the oral cavity.

Exclusion Criteria:

* Patients who are allergic to honey products.
* Patients on HRT (hormone replacement therapy) or patients who have not had a menstrual cycle for the last 12 months.
* Patients who had lost teeth because of periodontal disease.
* Patients who are or have been smokers in the past.
* Patients are on any kind of antibiotic therapy at the time of screening.
* Systemic conditions predispose patients to chronic periodontal diseases such as diabetes.

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — our participants comprises of peri-menopausal population so only the female candidates were selected.
Enrollment: 102 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Change in periodontal pocket depth. | baseline,6 weeks, 12 weeks.
  Measured in mm using calibrated williams periodontal probe.
Change in clinical attachment loss. | baseline,6 weeks, 12 weeks
  Measured in mm using calibrated williams periodontal probe.
change in Bleeding on probing. | baseline,6 weeks, 12 weeks
  Presence or absence of blood in gingival pockets on probing.

SECONDARY OUTCOMES:
Change in salivary neopterin levels. | baseline and 12 weeks.
  Saliva samples were taken and stored before and after the treatment to check the levels of Neopterin through Elisa.

CONTACTS AND LOCATIONS:
Overall Officials: Syeda M. Waqar, M.Phil, Principal Investigator — Ziauddin University, shahrae ghalib, Clifton, Karachi. Pakistan.
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
it was written in the consent form that no information regarding patients will be shared to anyone in any case considering the ethics.

REFERENCES:
- [Background] Waqar SM, Huma A, Razi A, Saher F, Qureshi SS, Qureshi JA. FORMULATION DEVELOPMENT AND EVALUATION OF PROPOLIS MOUTHWASH FOR TREATMENT OF PERIODONTAL DISEASE.
- [Derived] Waqar SM, Razi A, Qureshi SS, Saher F, Zaidi SJA, Kumar C. Comparative evaluation of propolis mouthwash with 0.2% chlorhexidine mouthwash as an adjunct to mechanical therapy in improving the periodontitis among perimenopausal women: a randomized controlled trial. BMC Oral Health. 2024 Jan 5;24(1):26. doi: 10.1186/s12903-023-03768-4. PMID 38183081